CLINICAL TRIAL: NCT06571110
Title: Analgesic Response to Opioids in Patients With Fibromyalgia After Conventional Acupuncture Versus Sham Acupuncture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Ariana M. Nelson, MD, Associate Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4736
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia
Keywords: Acupunture
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional acupuncture (Active Comparator): During TA, 9 acupuncture needles (Seirin 0.25 · 50 mm) are inserted at GV20,earShenmen,LI4,LI11,SP6,LR3,GB34,and bilateral ST 36. Needle insertion depth is approximately 2 cm for all TA points except for DU 20 and ear Shenmen, which have shallower insertion depths. All needles below the neck level are manually manipulated to elicit De Qi sensations.
  Interventions: Procedure: Traditional Acupuncture
- Sham acupuncture (Sham Comparator): SA participants experience a non-skin penetrating pricking sensation at 9 non-acupuncture point locations, sham intervention did not penetrate the skin and was designed to not elicit De Qi. somatosensory component generated by this procedure would be likely to be less than the skin penetrating-TA protocol that elicited De Qi. The sham locations were within similar body locations as the TA points; however, the SA location is not on known acupuncture points or meridians.
  Interventions: Procedure: Sham Acupuncture

INTERVENTIONS:
Procedure: Traditional Acupuncture — Acupuncture is a type of treatment where thin needles are gently inserted into specific parts of your body. It's often used to help with things like pain, headaches, stress, and anxiety.
  Arms: Traditional acupuncture
Procedure: Sham Acupuncture — Sham acupuncture in this trial involves the insertion superficially to mimic the procedure of true acupuncture without providing any therapeutic effect. The needles will be similar to those used in the true acupuncture group but will not be stimulated, ensuring blinding and controlling for placebo effects.
  Arms: Sham acupuncture

SUMMARY:
This study aims to see whether acupuncture can help fibromyalgia patients by giving them acupuncture treatment and seeing whether acupuncture helps enhance the effects of an opioid.

DETAILED DESCRIPTION:
The investigator hypothesizes that traditional acupuncture (TA) enhances binding of the MOR receptor which will then enhance the pain-reducing effects of opioids compared to sham acupuncture (SA). The investigator will test the hypothesis by giving participants a validated Brief Pain Inventory to complete during the pre-therapy opioid challenge and one week after TA or SA therapy is completed.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 - 80 years old
* have been diagnosed with Fibromyalgia for more than 6 months
* Are already using chronic, continuous opioid therapy, including but not limited to the use of Hydrocodone (Norco), Oxycodone (Percocet), morphine, methadone or Tylenol #3 daily
* Have moderate to excruciating pain at baseline, determined by a 5 or greater score on the Visual Analogue Scale (VAS)

Exclusion Criteria:

* Are younger than 18 or older than 80 years old
* Have been diagnosed with a Substance Use Disorder (SUD)
* Pregnant
* Have an active litigation or worker's compensation case
* Have an active mental health diagnosis, such as bipolar disorder, psychosis, or suicidal ideation
* Are prescribed and actively using low dose Naltrexone . Have tried acupuncture in the last 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the pain VAS versus time following opioid challenge for pre-post TA vs. pre-post SA | Change in pain score after opioid administration comparing the first and last study treatment session (2 weeks separation in time).
  We hypothesize that patients randomized to TA treatment will have a statistically greater change in pain after the final opioid challenge compared to the initial opioid challenge, as compared to patients randomized to SA treatment(p-value set at 0.05).

SECONDARY OUTCOMES:
Change in FIQ | Change in pain score after opioid administration comparing the first and last study treatment session (2 weeks separation in time).
  patients' response to pain interference over the past 7 days as assessed by the Fibromyalgia Impact Questionnaire in both patient groups to ensure a similar response to TA and SA as reflected in prior studies. The minimum value is: 0 and the maximum value is: 100. A Higher score on the FIQ indicates a worse outcome, meaning greater impact of fibromyalgia on the individual's daily life and overall functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Ariana Nelson, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Health Susan Samueli Integrative Health Institute, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mawla I, Ichesco E, Zollner HJ, Edden RAE, Chenevert T, Buchtel H, Bretz MD, Sloan H, Kaplan CM, Harte SE, Mashour GA, Clauw DJ, Napadow V, Harris RE. Greater Somatosensory Afference With Acupuncture Increases Primary Somatosensory Connectivity and Alleviates Fibromyalgia Pain via Insular gamma-Aminobutyric Acid: A Randomized Neuroimaging Trial. Arthritis Rheumatol. 2021 Jul;73(7):1318-1328. doi: 10.1002/art.41620. Epub 2021 May 31. PMID 33314799
- [Background] Zucker NA, Tsodikov A, Mist SD, Cina S, Napadow V, Harris RE. Evoked Pressure Pain Sensitivity Is Associated with Differential Analgesic Response to Verum and Sham Acupuncture in Fibromyalgia. Pain Med. 2017 Aug 1;18(8):1582-1592. doi: 10.1093/pm/pnx001. PMID 28340147
- [Background] Harris RE, Clauw DJ, Scott DJ, McLean SA, Gracely RH, Zubieta JK. Decreased central mu-opioid receptor availability in fibromyalgia. J Neurosci. 2007 Sep 12;27(37):10000-6. doi: 10.1523/JNEUROSCI.2849-07.2007. PMID 17855614
- [Background] Murphy AE, Buchtel H, Mawla I, Ichesco E, Larkin T, Harte SE, Zhan E, Napadow V, Harris RE. Temporal Summation but Not Expectations of Pain Relief Predict Response to Acupuncture Treatment in Fibromyalgia. J Pain. 2024 Oct;25(10):104622. doi: 10.1016/j.jpain.2024.104622. Epub 2024 Jul 8. PMID 38986891
- [Background] Harris RE, Tian X, Williams DA, Tian TX, Cupps TR, Petzke F, Groner KH, Biswas P, Gracely RH, Clauw DJ. Treatment of fibromyalgia with formula acupuncture: investigation of needle placement, needle stimulation, and treatment frequency. J Altern Complement Med. 2005 Aug;11(4):663-71. doi: 10.1089/acm.2005.11.663. PMID 16131290
- [Background] Schrepf A, Harper DE, Harte SE, Wang H, Ichesco E, Hampson JP, Zubieta JK, Clauw DJ, Harris RE. Endogenous opioidergic dysregulation of pain in fibromyalgia: a PET and fMRI study. Pain. 2016 Oct;157(10):2217-2225. doi: 10.1097/j.pain.0000000000000633. PMID 27420606
- [Background] Harte SE, Clauw DJ, Napadow V, Harris RE. Pressure Pain Sensitivity and Insular Combined Glutamate and Glutamine (Glx) Are Associated with Subsequent Clinical Response to Sham But Not Traditional Acupuncture in Patients Who Have Chronic Pain. Med Acupunct. 2013 Apr;25(2):154-160. doi: 10.1089/acu.2013.0965. PMID 24761170
- See also: Greater Somatosensory Afference With Acupuncture Increases Primary Somatosensory Connectivity and Alleviates Fibromyalgia Pain via Insular γ-Aminobutyric Acid: A Randomized Neuroimaging Trial — https://www.ncbi.nlm.nih.gov/pmc/articles/pmid/33314799/
- See also: Evoked Pressure Pain Sensitivity Is Associated with Differential Analgesic Response to Verum and Sham Acupuncture in Fibromyalgia — https://www.ncbi.nlm.nih.gov/pmc/articles/pmid/28340147/
- See also: Decreased central mu-opioid receptor availability in fibromyalgia — https://www.ncbi.nlm.nih.gov/pmc/articles/pmid/17855614/
- See also: Temporal Summation but Not Expectations of Pain Relief Predict Response to Acupuncture Treatment in Fibromyalgia — https://linkinghub.elsevier.com/retrieve/pii/S1526-5900(24)00563-7
- See also: Endogenous opioidergic dysregulation of pain in fibromyalgia: a PET and fMRI study — https://www.ncbi.nlm.nih.gov/pmc/articles/pmid/27420606/
- See also: Pressure Pain Sensitivity and Insular Combined Glutamate and Glutamine (Glx) Are Associated with Subsequent Clinical Response to Sham But Not Traditional Acupuncture in Patients Who Have Chronic Pain — https://www.ncbi.nlm.nih.gov/pmc/articles/pmid/24761170/